CLINICAL TRIAL: NCT04511052
Title: Probiotics for Enhanced Tissue Carotenoid Status: a Double-blind, Randomized, Controlled Trial
Brief Title: Probiotics for Enhanced Tissue Carotenoid Status in Premenopausal Women
Acronym: ProCar
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Principal Investigator, Stan Kubow, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A12-M57-19B; IT15250 (Other Grant/Funding Number: MITACS Accelerate)
Record Dates: First submitted 2020-07-29; First posted 2020-08-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Carotenoid Status; Gut Microbiome; Skin Health
Keywords: Carotenoid; Microbiome; Skin; Color; Plasma
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carotenoid + Probiotic (Experimental): Carotenoid: 1 capsule daily of a mixed carotenoid (~ 20 mg total carotenoids) supplement
  Probiotic: 1 capsule daily containing 10 x 10^9 CFU of a proprietary strain
  Total duration: 10 weeks
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Carotenoid supplement
- Carotenoid + Placebo (Placebo Comparator): Carotenoid: 1 capsule daily of a mixed carotenoid (~ 20 mg total carotenoids) supplement
  Placebo: 1 capsule daily containing the same carrier material of the probiotic, that is also similar in size, shape, and taste.
  Total duration: 10 weeks
  Interventions: Other: Placebo; Dietary Supplement: Carotenoid supplement

INTERVENTIONS:
Dietary Supplement: Probiotic — Daily intake of 10 x 10^9 CFU of a proprietary strain for a total duration of 10 weeks
  Arms: Carotenoid + Probiotic
Other: Placebo — 1 capsule daily containing the same carrier material that is similar in size, shape and taste to the probiotic, for a duration of 10 weeks
  Arms: Carotenoid + Placebo
Dietary Supplement: Carotenoid supplement — 1 capsule daily containing ~20 mg of total carotenoids for a total duration of 10 weeks

SUMMARY:
Carotenoids are yellow-orange fat soluble plant pigments primarily obtained from the diet that serve as an accurate biomarker for fruit and vegetable intake. Carotenoids have demonstrated antioxidant, anti-inflammatory, and anti-obesogenic properties among others. Excess carotenoids are deposited in the skin for storage where they protect against UV skin damage and contribute to improvements in skin health (i.e., decrease the appearance of wrinkles). However, carotenoid status is linked to bioavailability and absorption, which has a high inter-individual variability. It has been hypothesized that inter-individual variations are related to the diversity of gut microbiota.

The aim of the present study is to determine whether probiotic supplementation can enhance carotenoid status and responsiveness to carotenoid-mediated changes in blood and skin from intake of a supplement containing mixed forms of carotenoids in pre-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-menopausal or non-perimenopausal women,
2. 30-50 years of age,
3. BMI of 18.5 - 29.9 kg/m2,
4. Access to a smartphone that has a camera and iOS 11.0 or Android 4.2 and up,
5. Visible fine to moderate wrinkles on the face (e.g. forehead, crow's feet area, etc.),
6. Fitzpatrick scale of types I, II, & III
7. Urine pregnancy test of negative
8. Willing to maintain current physical activity and dietary habits
9. Willing to refrain from taking natural health products containing carotenoids (beta-carotene, lutein, lycopene, etc.)
10. Willing to discontinue consumption of probiotic supplements and food containing added probiotics (e.g. yogurts with live, active cultures or supplements) or fermented foods (e.g. Kefir, pickles, etc.) upon screening and for the duration of the study,
11. Willing to apply the moisturizer provided on every day throughout the study upon admission to the study (about -2 weeks),
12. Willing to refrain from using any cream (including the moisturizer provided) and makeup on the face for study visits and photo capture (face, eyes and lips),
13. Able to understand and comply with requirements of the study (e.g. complete all clinical visits, questionnaires, records, and diaries),
14. Able to provide a written informed consent.

Exclusion Criteria:

1. Known immunodeficiency (immuno-compromised and immuno-suppressed participant; e.g. AIDS, lymphoma, participants undergoing long-term corticosteroid treatment, chemotherapy and allograft participant),
2. Known chronic or acute illness (e.g. hepatitis, diabetes, high blood pressure, jaundice, etc.), unless under control via medication,
3. History of illness or use of any type of drug that may interfere with the investigational product or intervention (e.g. antibiotics) within 1 month of screening (may be eligible to participate after a 2-week washout period),
4. Known chronic or acute skin condition on the face (e.g. eczema, psoriasis, severe acne, rosacea, etc.),
5. Facial surgery (e.g. lifting, facial rejuvenation) or chemical treatment (e.g. Botox injection) within 5 years before study start,
6. Frequent tanning salons, use tanning products, or foresee high exposure to the sun during the study,
7. Tattoos on the face or palms of the hands,
8. Milk, soy or yeast allergy,
9. Routine use of dietary supplements that may interfere with outcomes measured (e.g. anti-oxidant, anti-inflammatory, herbal),
10. Use of probiotic products in the past 2 weeks (may be eligible to participate after a 2-week washout period),
11. Allergy to any of the ingredients contained in the moisturizer provided,
12. Use of antiaging creams containing retinol, glycolic acid, Coenzyme Q, etc. (may be eligible to participate after a 2 weeks washout period upon admission to the study),
13. Current smoker (tobacco or cannabis),
14. Excessive alcohol consumption (>1 drink/day),
15. Drug abuse or addiction,
16. Bleeding/blood disorder
17. Psychological disorder
18. Currently enrolled in another trial
19. Positive pregnancy test in women of child-bearing potential; breast-feeding or planning on becoming pregnant during the course of the study (determined by a pregnancy test performed at the screening visit),
20. Women of child-bearing potential not using effective contraception which include:

    * Hormonal contraceptives including combined oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormonal implants
    * Intrauterine devices (IUD) or Intrauterine system (IUS)
    * Tubal ligation
    * Vasectomy of partner
    * Barrier method (condom or occlusive cap with spermicide)
    * Abstinence
21. Participation in a similar study within 3 months of the screening visit.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Changes in skin yellow color saturation measured by a spectrophotometer | Week 0, 5, and 10
  Average b* value (yellow coloration designated by the CIELab color space) measured from the palm and forehead by spectrophotometry

SECONDARY OUTCOMES:
Changes in blood plasma carotenoid status | Week 0, 5, and 10
  Blood plasma HPLC or LC-MS analysis
Changes in yellow skin color saturation measured by image analysis | Week 0, 5, and 10
  Average b* value (yellow coloration designated by the CIELab color space) measured by image analysis of the palm and forehead
Changes in fecal microbial composition | Week -2, 0, 5, and 10
  16s rRNA sequencing
Changes in recovery of probiotic strain | Week -2, 0, 5, and 10
  16s rRNA qPCR
Changes in skin hydration | Week 0, 5, and 10
  Measured using a Courage + Khazaka probe system
Changes in skin elasticity | Week 0, 5, and 10
  Measured using the Tewameter probe from Courage + Khazaka probe system
Changes in skin trans-epidermal water loss | Week 0, 5, and 10
  Measured using a Courage + Khazaka probe system
Changes in facial skin wrinkling | Week 0, 5, and 10
  Images of participants will be individually rated by two trained specialists based on the skin aging atlas 1 - Caucasian type book at four different regions: forehead, crow's feet, nasolabial fold, and upper lip
Changes in plasma interleukin 1β (IL-1β) levels | Week 0, 5, and 10
  Assessed with MILLIPLEX MAP Human High Sensitivity T Cell Panel - Immunology Multiplex Assay.
Changes in plasma interleukin-6 (IL-6) levels | Week 0, 5, and 10
  Assessed with MILLIPLEX MAP Human High Sensitivity T Cell Panel - Immunology Multiplex Assay.
Changes in plasma interleukin-8 (IL-8) levels | Week 0, 5, and 10
  Assessed with MILLIPLEX MAP Human High Sensitivity T Cell Panel - Immunology Multiplex Assay
Changes in plasma tumor necrosis factor- α (TNF-α) levels | Week 0, 5, and 10
  Assessed with MILLIPLEX MAP Human High Sensitivity T Cell Panel - Immunology Multiplex Assay.
Changes in plasma 8-hydroxy-2'-deoxyguanosine (8-OHdG) levels | Week 0, 5, and 10
  Assessed via LC-MS
Changes in plasma F-2 isoprostane levels | Week 0, 5, and 10
  Assessed via LC-MS
Changes in plasma progesterone levels | Week 0, 5, and 10
  Analysis using MILLIPLEX MAP Multi-Species Hormone Magnetic Bead Panel
Changes in plasma estradiol levels | Week 0, 5, and 10
  Analysis using MILLIPLEX MAP Multi-Species Hormone Magnetic Bead Panel
Changes in plasma testosterone levels | Week 0, 5, and 10
  Analysis using MILLIPLEX MAP Multi-Species Hormone Magnetic Bead Panel
Changes in plasma cortisol levels | Week 0, 5, and 10
  Analysis using MILLIPLEX MAP Multi-Species Hormone Magnetic Bead Panel
Changes in plasma cholesterol levels | Week 0, 5, and 10
  Using a colorimetric assay
Changes in plasma antioxidant capacity | Week 0, 5, and 10
  Measured using the 2,2'-azino-bis-3-ethylbenzthiazoline-6-sulfonic acid (ABTS) assay
Changes in Vitamin A status | Week 0, 5, and 10
  Plasma HPLC analysis
Changes in perceived health and attractiveness | Week 0, 5, and 10
  A perception trial is a validated method used to determine the attractiveness preferences of participants (Lefevre & Perrett, 2015). Images of participants from the intervention trial will be sent to the Department of Psychology at McGill University, where the laboratory coordinator will set up an electronic survey that will display randomized sets of images from the same intervention participant at all timepoints (week 0, 5, and 10) of the intervention, in randomized order of presentation (left and right). A separate group of 60 participants will be recruited to participate in the perception trial and assess the images of the intervention participants. These participants will be trained using a few sample photos and then will be instructed to choose the most attractive and healthy looking face in a forced-choice paradigm for each comparison presented in the electronic survey.
Changes in quality of life assessed by SF-36 questionnaire | Week 0, 5, and 10
  The short form 36-Item Health Survey 1.0 Questionnaire is a validated questionnaire that will be used to assess QoL as a recent study (Valler-Colomer et al., 2019) demonstrated a consistent association between higher QoL indicators and particular gut microbiota profiles (butyrate-producing Faecalibacterium and Coprococcus bacteria). This survey consists of 36 items that average together to indicate eight scale scores for various health indicators (e.g., emotional well-being, general health, etc.). Scores range from 0-100, with higher scores representing better health. Carotenoid supplementation has also demonstrated improvements in sub-optimal symptoms of physical and emotional health measured via various self-reported questionnaires (Stringham et al., 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Emily Clinical Nutrition Research Unit (7 rue maple), Sainte-Anne-de-Bellevue, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No